CLINICAL TRIAL: NCT01747369
Title: Surveillance of Hospitalised Pneumonia and Bacterial Meningitis in Tône District, Togo, 2010-2013
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Agence de Médecine Préventive, France (Other)
Collaborators: Region Sanitaire des Savanes, Togo (Unknown); Ministere de la Sante et de la Promotion Sociale, Togo (Unknown); Institut National d'Hygiene, Togo (Unknown); Centre Muraz (Other); Fondation Mérieux, France (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: PneumoTone
Record Dates: First submitted 2011-07-04; First posted 2012-12-11 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Pneumonia, Bacterial; Pneumonia, Viral; Meningitis, Bacterial
Keywords: surveillance study; prospective; observational; health center-based; pneumonia, bacterial; pneumonia, viral; meningitis, bacterial; Africa south of the Sahara
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia, Viral; Meningitis, Bacterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, cerebro-spinal fluid, nasal aspirate
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to estimate the burden of disease due to pneumococci, other bacteria and viruses in the African meningitis belt prior to pneumococcal conjugate vaccine introduction and to estimate the population impact of the vaccine after its implementation in 2014. In a defined population of a sanitary district in northern Togo, during the period 2010 to 2017, investigators enroll patients of all ages with suspected pneumonia requiring hospitalization or suspected bacterial meningitis. Patients are evaluated by bacteriology and molecular biology techniques on blood, cerebro-spinal fluid, nasal aspirates and by chest X-ray.

ELIGIBILITY:
Pneumonia surveillance:

Inclusion Criteria:

* resident of Tône sanitary district - requiring hospitalisation for at least one night for clinical pneumonia syndrome
* hospitalised in a study site during the study period

Exclusion Criteria:

* absence of informed consent by patient or legal tutor

Meningitis surveillance:

Inclusion Criteria:

* resident of Tône sanitary district
* presenting clinical signs of acute bacterial meningitis
* hospitalised in a study site during the study period

Exclusion Criteria:

* absence of informed consent by patient or legal tutor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pneumonia surveillance:
  -residents of Tône sanitary district requiring hospitaliation for suspected pneumonia and presenting at one of the hospitals of Dapaong town (district capital)
  Meningitis surveillance:
  - residents fo Tône sanitary district presenting with suspected meningitis at one of the hospitals of Dapaong town (district capital) or Sinkasse health center
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumococcal pneumonia requiring hospitalisation, confirmed by blood culture or PCR analysis of blood | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)
Incidence of pneumococcal meningitis, confirmed by culture or PCR on cerebro-spinal fluid | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)

SECONDARY OUTCOMES:
Incidence of radiologically confirmed pneumonia requiring hospitalisation | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)
Incidence of suspected pneumonia requiring hospitalisation with elevated C-reactive protein serum concentration (<40mg/l) | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)
Incidence of suspected pneumonia requiring hospitalisation with reduced oxygen saturation (<90%) | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)
Incidence of pneumonia of other bacterial or viral etiology requiring hospitalisation | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)
Incidence of acute meningitis of other bacterial etiology | Subjects will be enrolled on admission to hospital and followed for the duration of hospitalization (median duration 6 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Moïsi, PhD, Principal Investigator — Agence de Médecine Préventive
Locations (5):
- Togo (5):
  - Centre Hospitalier Régional (CHR) Savanes, Dapaong, Savanes
  - Clinique Win' Pang, Dapaong, Savanes
  - Hôpital d'enfants Yendubé, Dapaong, Savanes
  - Polyclinique, Dapaong, Savanes
  - Centre médico-social (CMS), Sinkassé, Savanes